CLINICAL TRIAL: NCT06937359
Title: Prospective Observational Study of Self-Reported Outcomes in Reiki Healing in the Netherlands Using the Measure Yourself Medical Outcomes Profile (MYMOP)
Brief Title: Healing Space Reiki Therapy: Effectiveness and Experiences
Status: Completed | Type: Observational
Sponsor: Louis Bolk Institute (Other)
Collaborators: Healing Space (Unknown); National Research Centre of Complementary and Alternative Medicine, Norway (Other)
Responsible Party: Principal Investigator, Herman van Wietmarschen, PhD, Louis Bolk Institute
Other Study IDs: 2025HSR
Record Dates: First submitted 2025-04-09; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: The Focus of the Study is on Any Volunteer With Any Symptom or Condition
Keywords: Reiki; MYMOP; symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reiki healing — Each client received four treatments with Healing Space Reiki Therapy: a foundation of Reiki, combined with a fully customized treatment with trauma processing and adjustments in diet and lifestyle at Dojo In Reiki treatments. In the Dojo In, there were 8 futons, with two Reiki Therapists at each futon treating one client. During these sessions, participants receive 4 Reiki treatments, each lasting about an hour, over 4 consecutive weeks. During these days, 2 trained and/or still training Reiki Therapists per treatment table provide a Reiki treatment under the supervision of the founders of Healing Space.
  Other Names: energy healing; biofield therapy

SUMMARY:
Reiki is an energetic healing method in which a therapist uses his hands on or near the clients body to channel life energy and send it to the client. This activates healing within the client and restores balance.

In this study clients at the Reiki training institute Healing Space are monitored for 4 weeks during 4 weekly Reiki healing sessions. Any client 18 years or older with any complaint can participate. A validated MYMOP questionnaire is used to monitor one main complaint, one secondary complaint and overall wellbeing after each of the 4 treatment sessions and before the start of treatment. A small number of clients will be interviewed for additional in depth data about their experiences. The aim of the study is to gain understanding about the effectiveness of Reiki.

DETAILED DESCRIPTION:
Given the substantial international socio-economic burden of healthcare, the development of inexpensive, safe, and evidence-based treatments is highly desirable. Reiki, as a non-invasive and low-cost therapy, holds potential as a complementary approach to conventional medical treatments. However, the lack of consensus on its efficacy and mechanisms necessitates further investigation. This study aims to address these gaps by exploring the conditions clients report when visiting a Reiki healer and evaluating the subjective effectiveness and experiences of Reiki therapy. By doing so, the study seeks to contribute to the growing body of evidence on Reiki and inform its potential integration into healthcare systems.

This study is an observational prospective pre-post study with a convenience sample. The study is conducted at the Healing Space Reiki center in the Netherlands by Reiki practitioners trained at Healing Space. Each Reiki session lasts 1 hour and is conducted by 2 Reiki practitioners supervised by the founders of Healing Space. MYMOP questionnaires are provided before the first treatment (baseline) and then after each of the 4 treatments. A number of interviews is conducted after the complete treatment. All participants provided written informed consent. A waiver for full ethical assessment will be obtained from an ethical committee.

The MYMOP complaints are categorized into four primary groups: pain, psychological problems, fatigue, and other. Pre- and post comparisons of the four MYMOP measurements were performed usign paired t-tests and independent sample t-tests. Interviews are analysed thematically.

ELIGIBILITY:
Inclusion Criteria:

* Presence of any self reported complaint
* 18 years or older
* No other treatments for this complaint during the intervention period

Exclusion Criteria:

* Other treatments for the complaint during the intervention period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult person with any complaint contacting Healing Space for treatment
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Self reported main symptom | 1 week
  Self reported main symptom measured with the MYMOP questionnaire.

SECONDARY OUTCOMES:
Self reported secondary symptom | 1 week
  Self reported secondary symptom with the MYMOP questionnaire
Overall wellbeing | 1 week
  Self reported overall welbeing with the MYMOP questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Healing Space, Bussum, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized MYMOP data and demographic data
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: September 2024 till end of 2026
Access Criteria: NAFKAM will access anonymized MYMOP and demographic data in excel format